CLINICAL TRIAL: NCT02318043
Title: Is Adenosine Monophosphate Superior to Histamine for Bronchial Provocation Test in Evaluation of Asthma?
Brief Title: AMP-BPT and His-BPT for Assessment of Asthma
Acronym: AMPHis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Jinping Zheng, Professor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: GWJ
Record Dates: First submitted 2014-12-07; First posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Asthma
Keywords: adenosine monophosphate; histamine; bronchial provocation test; asthma symptom score; asthma control
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMP-BPT (Active Comparator): Methods of AMP-BPT, by applying dosimeters, resembled that reported previously [see references 21-25]. Briefly, dilutions were delivered via nebulizers (output: 160 μl/min) using automated APS pro system (JAEGER, Hochburg, Germany). Inhalation challenge with normal saline served as control step. Challenge steps were proceeded if FEV1 fall <15% and restored to <10% within 1 minute. Subsequent inhalation challenges were performed at 1-minute intervals, and ceased when FEV1 fell by ≥20%. Salbutamol was administered via spacer (Volumatic, Allen & Hanbury's, UK). Spirometry was reexamined at minutes 3, 5, 10 and thereafter, to ensure safety, before discharge.
  Interventions: Drug: inhaled corticosteroids (usually budesonide/fomorterol 160/4.5mcg; fluticasone/salmeterol 250/50mcg)
- His-BPT (Active Comparator): Methods of His-BPT, by applying dosimeters, resembled that reported previously [see references 21-25]. Briefly, dilutions were delivered via nebulizers (output: 160 μl/min) using automated APS pro system (JAEGER, Hochburg, Germany). Inhalation challenge with normal saline served as control step. Challenge steps were proceeded if FEV1 fall <15% and restored to <10% within 1 minute. Subsequent inhalation challenges were performed at 1-minute intervals, and ceased when FEV1 fell by ≥20%. Salbutamol was administered via spacer (Volumatic, Allen & Hanbury's, UK). Spirometry was reexamined at minutes 3, 5, 10 and thereafter, to ensure safety, before discharge.
  Interventions: Drug: inhaled corticosteroids (usually budesonide/fomorterol 160/4.5mcg; fluticasone/salmeterol 250/50mcg)

INTERVENTIONS:
Drug: inhaled corticosteroids (usually budesonide/fomorterol 160/4.5mcg; fluticasone/salmeterol 250/50mcg) — Patients with uncontrolled and partly controlled asthma, following accomplishment of study 1, were invited to participate in observational study (study 2), which sought to determine usefulness of both BPTs in reflecting improvement of asthmatic symptoms following 3 and 6 months of moderate-dose ICSs treatment (400~800μg budesonide or equivalent). Patient continued to administer their original ICS during follow-up. During two follow-up visits (3 months apart), AMP-BPT, His-BPT and Hogg's symptom scores were reassessed.

SUMMARY:
Adenosine monophosphate (AMP) may reflect airway inflammation and hyperresponsiveness, but relationship between AMP and histamine (His, a conventional stimulus) bronchial provocation test (BPT) in asthma is not fully elucidated.

The investigators aimed to compare both BPTs and determine their usefulness in reflecting changes of asthmatic symptoms.

BPTs were performed in cross-over fashion, at 2-4day intervals. Cumulative doses eliciting 20% FEV1fall (PD20FEV1), diagnostic performance and adverse events were compared. Patients with PD20FEV1 lower than geometric mean were defined as responders, otherwise poor responders. Patients with uncontrolled and partly controlled asthma, who maintained their original inhaled corticosteroids therapy, underwent reassessment of airway responsiveness and asthmatic symptoms 3 and 6 months after.

DETAILED DESCRIPTION:
Airway hyperresponsiveness, the pivotal feature of asthma, can be assessed by bronchial provocation tests (BPTs), which may elicit bronchoconstriction via inhalation of stimuli. Histamine has been a direct stimulus for inducing bronchoconstriction via vasodilation, eosinophil chemotaxis and tissue edema. Clinically, histamine BPT (His-BPT) has gained extensive application for decades owing to the assay sensitivity and feasibility, but could not ideally predict anti-inflammatory treatment outcomes in practice. Additionally, mild adverse events (flushing and hoarseness) and insufficient capacity of identifying exercise-induced asthma have hampered further clinical applications.

Adenosine monophosphate (AMP) is an inflammatory mediator that serves as an indirect bronchial stimulus for detecting airway hyperresponsiveness in asthma. Compared with histamine, AMP may be pathophysiologically more relevant to airway inflammation and hyperresponsiveness and has been linked to presence and magnitude of atopy. However, differences of response to AMP-BPT and His-BPT in different asthma control levels and their associations with asthmatic symptom scores have not been fully elucidated.

We hypothesized that asthmatic patients, regardless of control levels, responded differentially to AMP-BPT and His-BPT, and that greater reduction in airway responsiveness to AMP (esp. responders of AMP-BPT) was associated with significant symptom alleviation. Henceforth, we sought to: 1) compare diagnostic performance and safety of AMP-BPT and His-BPT in different asthma control levels; 2) determine the association between airway responsiveness and asthmatic symptom scores.

Currently, His-BPT is recommended by the Chinese guideline and shares considerable similarity with methacholine (another conventional stimulus) BPT, we therefore did not perform the latter in this study.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18~65 years;
2. nil respiratory infection within 3 weeks;
3. normal chest radiography;
4. baseline FEV1>60% predicted;
5. withdrawn from, if any, oral leukotriene modifiers, corticosteroid or anti-histamine for 5 days, oral xanthenes or long-acting bronchodilators for 2 days, inhaled corticosteroids (ICSs) for 24 hours, and salbutamol for 6 hours

Exclusion Criteria:

1. FEV1 fall ≥20% following saline inhalation;
2. other chronic lower respiratory diseases (i.e. COPD);
3. severe systemic diseases (i.e. uncontrolled hypertension, malignancy);
4. limited understanding.

For healthy subjects, they had to be aged 18~65 years and had nil respiratory infection within 3 weeks, systemic diseases and had normal lung function.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cumulative dose eliciting 20% fall in FEV1 (PD20FEV1) | up to 12 months (Jan 2007 to Dec 2007)
  Cumulative dose eliciting 20% fall in FEV1 (PD20FEV1), reported as
Asthma symptom score as proposed by Hoggs et al | up to 12 months (Jan 2007 to Dec 2007)
  Asthma symptom score recorded within 1 week, with the highest possible score of 42 for the whole week

SECONDARY OUTCOMES:
Baseline spirometry (FVC, FEV1, FEV1/FVC, MMEF, PEF) | up to 12 months (Jan 2007 to Dec 2007)
  FVC, FEV1, FEV1/FVC, MMEF, PEF
Maximal decrease in FVC following bronchial provocation (expressed as percentage) | up to 12 months (Jan 2007 to Dec 2007)
  Maximal decrease in FVC following bronchial provocation, expressed as percentage as compared with baseline levels
Maximal decrease in FEV1 following bronchial provocation (expressed as percentage) | up to 12 months (Jan 2007 to Dec 2007)
  Maximal decrease in FEV1 following bronchial provocation, expressed as percentage as compared with baseline levels
Maximal decrease in MMEF following bronchial provocation (expressed as percentage) | up to 12 months (Jan 2007 to Dec 2007)
  Maximal decrease in MMEF following bronchial provocation, expressed as percentage as compared with baseline levels
Maximal decrease in PEF following bronchial provocation (expressed as percentage) | up to 12 months (Jan 2007 to Dec 2007)
  Maximal decrease in PEF following bronchial provocation, expressed as percentage as compared with baseline levels
Assay positivity of AMP-BPT and His-BPT (expressed as percentage) | up to 12 months (Jan 2007 to Dec 2007)
  Assay positivity of AMP-BPT and His-BPT, expressed as percentage
Diagnostic performance of AMP-BPT and His-BPT (area under the receiver operation characteristic curve, sensitivity, specificity, Youden index) | up to 12 months (Jan 2007 to Dec 2007)
  area under the receiver operation characteristic curve, sensitivity, specificity, Youden index
Changes in post-treatment asthma symptom scores | up to 12 months (Jan 2007 to Dec 2007)
  post-treatment minus pre-treatment asthma symptom score
Changes in post-treatment PD20FEV1 | up to 12 months (Jan 2007 to Dec 2007)
  post-treatment minus pre-treatment PD20FEV1

OTHER OUTCOMES:
incidence of adverse events of both BPTs | up to 12 months (Jan 2007 to Dec 2007)
  adverse events of AMP-BPT and His-BPT

REFERENCES:
- [Background] O'Byrne PM, Inman MD. Airway hyperresponsiveness. Chest. 2003 Mar;123(3 Suppl):411S-6S. doi: 10.1378/chest.123.3_suppl.411s. PMID 12629006
- [Background] Hanania NA. Targeting airway inflammation in asthma: current and future therapies. Chest. 2008 Apr;133(4):989-98. doi: 10.1378/chest.07-0829. PMID 18398119
- [Background] Leuppi JD. Bronchoprovocation tests in asthma: direct versus indirect challenges. Curr Opin Pulm Med. 2014 Jan;20(1):31-6. doi: 10.1097/MCP.0000000000000009. PMID 24275928
- [Background] Janssens T, Verleden G, De Peuter S, Petersen S, Van den Bergh O. Predicting asthma treatment outcome at diagnosis: the role of symptom perception during a histamine challenge test. J Asthma. 2012 Apr;49(3):230-6. doi: 10.3109/02770903.2012.656864. Epub 2012 Feb 9. PMID 22316110
- [Background] Dor A, Liebhart J, Malolepszy J. [Comparison of exercise and histamine provocation tests in patients with bronchial asthma]. Pneumonol Alergol Pol. 1999;67(1-2):22-7. Polish. PMID 10481521
- [Background] Driver AG, Kukoly CA, Ali S, Mustafa SJ. Adenosine in bronchoalveolar lavage fluid in asthma. Am Rev Respir Dis. 1993 Jul;148(1):91-7. doi: 10.1164/ajrccm/148.1.91. PMID 8317821
- [Background] Ali S, Mustafa SJ, Driver AG, Metzger WJ. Release of adenosine in bronchoalveolar lavage fluid following allergen bronchial provocation in allergic rabbits. Am Rev Respir Dis 1991;143:A417
- [Background] Polosa R, Ng WH, Crimi N, Vancheri C, Holgate ST, Church MK, Mistretta A. Release of mast-cell-derived mediators after endobronchial adenosine challenge in asthma. Am J Respir Crit Care Med. 1995 Mar;151(3 Pt 1):624-9. doi: 10.1164/ajrccm/151.3_Pt_1.624. PMID 7881647
- [Background] van den Berge M, Kerstjens HA, Meijer RJ, de Reus DM, Koeter GH, Kauffman HF, Postma DS. Corticosteroid-induced improvement in the PC20 of adenosine monophosphate is more closely associated with reduction in airway inflammation than improvement in the PC20 of methacholine. Am J Respir Crit Care Med. 2001 Oct 1;164(7):1127-32. doi: 10.1164/ajrccm.164.7.2102135. PMID 11673197
- [Background] De Meer G, Heederik D, Postma DS. Bronchial responsiveness to adenosine 5'-monophosphate (AMP) and methacholine differ in their relationship with airway allergy and baseline FEV(1). Am J Respir Crit Care Med. 2002 Feb 1;165(3):327-31. doi: 10.1164/ajrccm.165.3.2104066. PMID 11818315
- [Background] Suh DI, Lee JK, Kim CK, Koh YY. Bronchial hyperresponsiveness to methacholine and adenosine 5'-monophosphate, and the presence and degree of atopy in young children with asthma. Clin Exp Allergy. 2011 Mar;41(3):338-45. doi: 10.1111/j.1365-2222.2010.03664.x. Epub 2011 Jan 24. PMID 21255136
- [Background] Suh DI, Lee JK, Kim CK, Koh YY. Methacholine and adenosine 5'-monophosphate (AMP) responsiveness, and the presence and degree of atopy in children with asthma. Pediatr Allergy Immunol. 2011 Feb;22(1 Pt 2):e101-6. doi: 10.1111/j.1399-3038.2010.01110.x. PMID 21342276
- [Background] Kim CK, Choi SJ, Lee JK, Suh DI, Koh YY. Bronchial hyperresponsiveness to methacholine and adenosine monophosphate and the degree of atopy in children with allergic rhinitis. Ann Allergy Asthma Immunol. 2011 Jan;106(1):36-41. doi: 10.1016/j.anai.2010.10.019. PMID 21195943
- [Background] The Respiratory Society of the Chinese Medical Association. Guidelines for lung function testing (Part 3): Histamine and methacholine bronchial provocation test. Zhonghua Jie He He Hu Xi Za Zhi 2014; 37:566-71
- [Background] O'Byrne P, Bateman ED, Bousquet JD. Global Initiative for Asthma (GINA). Global strategy for asthma management and prevention. Updated 2006. Available at http://www.ginasthma.org/Guidelines/guidelines-resources.html Latest accessed: Sep 20, 2014
- [Background] Hogg JC, James AL, Pare PD. Evidence for inflammation in asthma. Am Rev Respir Dis. 1991 Mar;143(3 Pt 2):S39-42. doi: 10.1164/ajrccm/143.3_Pt_2.S39. No abstract available. PMID 2003688
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Background] Brusasco V, Crapo R, Viegi G; American Thoracic Society; European Respiratory Society. Coming together: the ATS/ERS consensus on clinical pulmonary function testing. Eur Respir J. 2005 Jul;26(1):1-2. doi: 10.1183/09031936.05.00034205. No abstract available. PMID 15994380
- [Background] Zheng J, Zhong N. Normative values of pulmonary function testing in Chinese adults. Chin Med J (Engl). 2002 Jan;115(1):50-4. PMID 11930658
- [Background] Guan W, Zheng J, Gao Y, Jiang C, An J, Yu X, Liu W. Leukotriene D4 bronchial provocation test: methodology and diagnostic value. Curr Med Res Opin. 2012 May;28(5):797-803. doi: 10.1185/03007995.2012.678936. Epub 2012 May 3. PMID 22435894
- [Background] Guan W, Zheng J, Gao Y, Jiang C, Xie Y, An J, Yu X, Liu W, Zhong N. Leukotriene D4 and methacholine bronchial provocation tests for identifying leukotriene-responsiveness subtypes. J Allergy Clin Immunol. 2013 Feb;131(2):332-8.e1-4. doi: 10.1016/j.jaci.2012.08.020. Epub 2012 Oct 4. PMID 23040886
- [Background] Guan WJ, Zheng JP, Gao Y, Jiang CY, Shi X, Xie YQ, Liu QX, Jiang M, An JY, Yu XX, Liu WT, Zhong LP, Wu ZP, Zhong NS. Impulse oscillometry for leukotriene D4 inhalation challenge in asthma. Respir Care. 2013 Dec;58(12):2120-6. doi: 10.4187/respcare.02417. Epub 2013 May 28. PMID 23716710
- [Background] Guan WJ, Zheng JP, Gao Y, Jiang CY, Xie YQ, Shi X, Zhu Z, An JY, Yu XX, Liu WT, Zhong NS. Responsiveness to leukotriene D4 and methacholine for predicting efficacy of montelukast in asthma. J Thorac Dis. 2013 Jun;5(3):298-301. doi: 10.3978/j.issn.2072-1439.2013.02.01. PMID 23825762
- [Background] Guan WJ, Zheng JP, Shi X, Xie YQ, Jiang CY, Gao Y, Zhu Z, An JY, Yu XX, Liu WT. Response--dose ratio is a surrogate of cumulative provocative dosage for bronchial provocation tests in asthma. Lung. 2014 Oct;192(5):701-9. doi: 10.1007/s00408-014-9612-7. Epub 2014 Jun 24. PMID 24958577